CLINICAL TRIAL: NCT02893384
Title: Analgesic Effects of Local Anesthetic Serratus Plane Infiltration for Total Mastectomy Surgery: A Pilot Study
Brief Title: Local Anesthetic for Total Mastectomy Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-5729
Record Dates: First submitted 2016-08-05; First posted 2016-09-08 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Breast Pain
MeSH Terms: conditions — Mastodynia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Anesthetic Injection (Experimental): The intervention involves injection of local anesthetic (0.25% bupivacaine with 1:200,000 epinephrine) under direct vision in the serratus anterior muscle plane at the end of surgery.
  Local Anesthetic Injection above the serratus anterior
  Interventions: Drug: Local Anesthetic Injection above the serratus anterior
- Control Arm (No Intervention): Retrospective control group who have not had the new injection technique.

INTERVENTIONS:
Drug: Local Anesthetic Injection above the serratus anterior — This is a quantitative pilot study assessing whether a new technique of local anesthesia injection during mastectomy surgery gives better pain outcomes than the standard methods. Patients who meet inclusion criteria will be invited to partake and all patients will have the injection technique. These patients will then be monitored for pain outcomes up to 7 days following the surgery and the results compared with historical results from patients who have already had the surgery.
  Other Names: Injection to serratus anterior muscle at the end of surgery
  Arms: Local Anesthetic Injection

SUMMARY:
Pain following mastectomy surgery for breast cancer can be significant. Poorly managed pain in the immediate time-period following surgery can potentially lead to long-term (chronic) pain conditions. There is still a need to find the safest, least invasive, and most effective method to manage this pain. The investigators believe that a new technique of injecting local anesthesia (freezing) in to specific areas at the end of mastectomy surgery may be a very important step to managing pain after breast surgery. The investigators would like to begin by performing a pilot study, meaning the investigators will perform the technique in patients and compare what their pain outcomes are to patients who have not had the technique.

DETAILED DESCRIPTION:
Mastectomy is associated with significant acute postoperative pain. It has been shown that inadequately managed post-mastectomy pain in breast cancer patients can have detrimental physiological, psycho-behavioural, recovery and healthcare utilization consequences. Most significantly, acute postoperative pain appears to be a substantial risk factor for progression to chronic post-surgical pain (CPSP), occurring in up to 68% of patients,, with higher severity of acute pain being linked with a greater progression to CPSP. A multimodal analgesic approach is the optimal method of reducing the risk of progression to CPSP, and there are a number of analgesic techniques that can be used to reduce the incidence of acute postoperative pain. Of the analgesic techniques used, the most common are multimodal systemic analgesia, thoracic paravertebral blockade, thoracic epidural analgesia, local anesthetic wound infiltration, and more recently pecs blocks and serratus plane blocks. The former three techniques are all associated with drawbacks including technical challenges, high risk of adverse effects, and limited evidence to minimize the progression to CPSP states, whilst local anesthetic wound infiltration has highly variable pain outcomes. Therefore, an alternative, safer, and more effective technique would be ideal.

Local infiltration analgesia (LIA) techniques have been demonstrated to be efficacious in joint surgery, whilst injection of local anesthesia in the serratus plane to target some of the intercostal and pectoral nerves may have some benefit in mastectomy surgery. However, nobody has yet performed LIA around these nerves in breast surgery, and the investigators feel that this has enormous potential.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective or urgent, primary, unilateral mastectomy with or without axillary lymph node dissection
* ASA-PS I-III
* 18-85 years of age, inclusive
* 50-100 kg, inclusive
* BMI 18 - 40

Exclusion Criteria:

* Bilateral mastectomy surgery
* Revision mastectomy surgery
* Inability or refusal to provide informed consent
* Chronic pain state
* Neuropathic pain
* Opioid dependence
* Allergy to local anesthesia
* Allergy to opioids

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-09; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in subjective Visual Analogue Scale (VAS) | 7 days after surgery
  The visual analogue scale is administered at different time points

SECONDARY OUTCOMES:
Patient Adverse Event Outcomes | 72 hours post operatively
  The visual analogue scale is administered at different time points

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Chan, MD, Principal Investigator — Toronto Western Hospital, University Health Network, University of Toronto

IPD SHARING:
Plan to Share IPD: Yes
publication